CLINICAL TRIAL: NCT01970592
Title: Skeletal Muscle Plasticity As An Indicator of Functional Performance Post-Stroke
Brief Title: Power Training Post-stroke
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: O0844-R
Record Dates: First submitted 2013-10-22; First posted 2013-10-28 (Estimated); Results first posted 2020-03-06 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2020-02

CONDITIONS: Stroke
Keywords: exercise; rehabilitation; walking
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- POWER (Experimental): Individuals with chronic post-stroke hemiparesis will undergo training to improve muscle power generation for 24 sessions (3 times/week) that includes both resistive and task-specific elements. Session duration will be ~90 minutes/day (inclusive of rest intervals). Training will include five distinct resistance activities aimed at improving muscle power-- each previously reported to contribute to improved walking.
  Interventions: Behavioral: POWER training

INTERVENTIONS:
Behavioral: POWER training — Individuals with chronic post-stroke hemiparesis will undergo training to improve muscle power generation for 24 sessions (3 times/week) that includes both resistive and task-specific elements. Session duration will be ~90 minutes/day (inclusive of rest intervals). Training will include five distinct resistance activities aimed at improving muscle power-- each previously reported to contribute to improved walking
  Other Names: strength training

SUMMARY:
Hemiparesis, strictly defined as (muscular) weakness affecting one side of the body, is seen in three-quarters of individuals following stroke. Weakness in this population results from both neural and muscular factors which include, respectively, the ability to activate skeletal muscle as well as the force generating capacity of the muscle. The overall goal is to improve walking in persons post-stroke by training subjects with an intervention that specifically targets existing neural and muscular impairments, thereby facilitating locomotor recovery.

DETAILED DESCRIPTION:
A primary impairment associated with post-stroke hemiparesis is the failure to make rapid graded adjustment of muscle force (i.e. muscle power) within the context of purposeful complex synergies (e.g., coordination during walking). Not surprisingly, the impact of stroke on walking is significant, with less than 50% of survivors progressing to independent community ambulation. Even among those who achieve independent ambulation, significant residual deficits persist in balance and gait speed, with ~75% of persons post-stroke reporting limitations in mobility related to walking. Muscle weakness is the most prominent motor consequence among the nearly 6 million survivors of stroke living in the United States and the strongest predictor of functional disability in this large clinical cohort. To date, the physiological mechanisms that contribute to muscle dysfunction in hemiparetic subjects are largely unstudied. Moreover, evidence regarding the efficacy of interventions aimed at attenuating impaired muscle function and the ensuing functional consequences in the post-stroke population is equivocal and viable therapeutic options to remediate hemiparetic muscle weakness remain among the most pressing challenges for biomedical research. The investigators propose that impaired muscle power (the product of muscle strength and velocity) generation is causal of functional (walking) disability post-stroke. In addition, coordination deficits are also critical determinants of functional performance. The investigators have developed a comprehensive theoretical framework that defines and measures the factors underlying disordered muscle function and coordination and will apply this framework to Post-stroke Optimization of Walking using Explosive Resistance (POWER) training. The investigators' goals over the four year funding period are to 1) quantify neural and muscular adaptations that contribute to impaired muscle power generation post-stroke; 2) assess effects of POWER training on neural and muscular adaptations in paretic and non-paretic muscle; and 3) determine the relationship between changes in neural and muscular adaptations following POWER training and locomotor improvements. Innovative aspects of the proposed work include the novel training intervention; the advanced magnetic resonance assessments; as well as the unique measure of the coordination that the investigators propose. It is the investigators' belief that: a) neural and muscular adaptations following stroke are associated with impaired muscle power generation as well as locomotor ability, b) POWER training attenuates functional deficits by addressing the underlying neural and muscular elements and c) functional improvements following training are predicated on improving the most prominent neural and muscular contributors to muscle power generation. If correct, the data generated will provide an entirely new level of evidence regarding the effectiveness of this novel intervention strategy on improving functional performance as well as the importance of peripheral muscle properties as predictors of locomotor ability post-stroke.

ELIGIBILITY:
Inclusion Criteria:

* age 50-70,
* stroke within the past 6 to 24 months,
* residual paresis in the lower extremity (Fugl-Meyer Lower Extremity motor score <34),
* ability to walk without assistance and without an ankle foot orthotic (AFO) on the treadmill 30 seconds at speeds ranging from 0.3 - 0.8 m/s, and
* provision of informed consent.
* In addition, all subjects who meet criteria for the training portion must complete an exercise tolerance test and be cleared for participation by the study cardiologist.

Exclusion Criteria:

* Unable to ambulate at least 150 feet prior to stroke, or experienced intermittent claudication while walking;
* rating on Modified Ashworth Scale 3 at the knee or ankle;
* limited lower extremity range of motion of the knee (passive flexion Range of Motion [ROM] < 90); hip (inability to achieve neutral 0 hip extension); or ankle (inability to achieve 0 of active dorsiflexion);
* history of congestive heart failure, unstable cardiac arrhythmias, hypertrophic cardiomyopathy, severe aortic stenosis, angina or dyspnea at rest or during activities of daily living (ADLs);
* History of chronic obstructive pulmonary disease (COPD) or oxygen dependence;
* Preexisting neurological disorders, dementia or previous stroke;
* History of major head trauma;
* Legal blindness or severe visual impairment;
* history of significant psychiatric illness
* Life expectancy <1 yr.,
* Severe arthritis or other problems that limit passive ROM;
* post-stroke depression (PHQ-9 10),
* History of deep vein thrombosis (DVT) or pulmonary embolism within 6 months;
* Uncontrolled diabetes with recent diabetic coma, or frequent insulin reactions;
* Severe hypertension with systolic >200 mmHg and diastolic >110 mmHg at rest;
* Previous or current enrollment in a trial to enhance motor recovery;
* Presence of non-magnetic resonance (MR) compatible implants, pregnancy or severe claustrophobia.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-10-01 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2019-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris M Gregory, PhD, Principal Investigator — Ralph H. Johnson VA Medical Center, Charleston, SC
Locations (1):
- Ralph H. Johnson VA Medical Center, Charleston, SC, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The pool of candidates were recruited from rehabilitation programs at the Medical University of South Carolina; the Ralph H. Johnson VAMC; and Charleston area communities.
Pre-assignment Details: After enrollment, participants were thoroughly evaluated for functional and cognitive impairments as well as physical performance. Descriptive physical performance testing included the lower extremity Fugl-Meyer Assessment (FMA-LE), Stroke Impact Scale (SIS), Berg Balance Scale (BBS) and the NIH Stroke Scale.
Period: Overall Study
Arm/Group | POWER
Started | 56 (Completed all training sessions)
Completed (Completed all training sessions) | 50
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | POWER
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants] — Age is self report or from medical records if available
  Participants
    <=18 years | 0
    Between 18 and 65 years | 44
    >=65 years | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (16.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 27
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 50
Self-selected walking speed [Mean (Standard Deviation); unit: meters per second] | 0.51 (0.29)
Maximum voluntary contraction [Mean (Standard Deviation); unit: foot pounds] | 62 (31)

OUTCOME MEASURES:

1. Primary Outcome: Gait Speed
Description: The speed the subject chooses to walk when instructed to walk at their "comfortable speed"
Time Frame: 8 weeks
Population: Individuals completing POWER training
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | POWER
Number analyzed (Participants) | 50
meters per second | 0.51 (0.29)

2. Secondary Outcome: Muscle Strength
Description: The strength of the paretic lower leg muscles will be measured by asking the participants to contract their muscles as forcefully as possible. Testing will be conducted on a specialized machine called an isokinetic dynamometer. This testing is designed to assess the ability to generate muscle power. Before testing the participants will be asked to perform 5 minutes of low intensity cycling. Strength testing will include movements at the hip, knee and ankle in both legs.
Time Frame: 8 weeks
Population: Individuals completing POWER training
Measure: Mean (Standard Deviation); unit: foot pounds
Arm/Group | POWER
Number analyzed (Participants) | 50
foot pounds | 62 (31)

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | POWER
All-Cause Mortality (participants affected / at risk) | 0/56
Serious Adverse Events (participants affected / at risk) | 1/56
Other Adverse Events (participants affected / at risk) | 3/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POWER (N=56)
Medical DIagnosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Lung cancer diagnosis
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | POWER (N=56)
Participant Fall (Musculoskeletal and connective tissue disorders) | 3 (56) — Minor injuries resulting from non-study related falls

LIMITATIONS AND CAVEATS:
None noted

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2011-07-14): https://cdn.clinicaltrials.gov/large-docs/92/NCT01970592/Prot_SAP_000.pdf